CLINICAL TRIAL: NCT01960842
Title: An Open-Label, Single-Arm, Baseline-Controlled, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of ABT-SLV187 Monotherapy in Subjects With Advanced Parkinson's Disease and Persistent Motor-Complications Despite Optimized Treatment With Available Anti-Parkinsonian Medication
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of ABT-SLV187 Monotherapy in Subjects With Advanced Parkinson's Disease (PD) and Persistent Motor Complications, Despite Optimized Treatment With Available Anti-Parkinsonian Medications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-921
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2016-04

CONDITIONS: Advanced Parkinson's Disease
Keywords: levodopa; Advanced Parkinson's Disease; carbidopa; levodopa-carbidopa intestinal gel; Safety and Efficacy
MeSH Terms: interventions — Jejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levodopa-Carbidopa Intestinal Gel (LCIG) (Experimental): All participants received LCIG via the N-J tube during the nasojejunal (N-J) Test Period and delivered to the proximal small intestine via percutaneous endoscopic gastrostomy - with jejunal extension tube (PEG-J) during the Post-PEG-J Long-Term Treatment Period. The starting dose was individually determined based on the daily dose of oral levodopa prior to study enrollment.
  The infusion dose was individually optimized for each participant on the basis of response and potential adverse events. During the PEG-J Period, LCIG was expected to be infused continuously over approximately 16 hours daily with a rate of infusion ranging from 1 to 10 mL/hour (20 to 200 mg of levodopa/hour).
  Interventions: Drug: Levodopa-carbidopa intestinal gel; Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: PEG tube; Device: J-tube

INTERVENTIONS:
Drug: Levodopa-carbidopa intestinal gel — Dose levels will be individually optimized. Infusion should be kept within a range of 0.5-10 mL/hour (10-200 mg levodopa/hour) and is usually 2-6 mL/hour (40-120 mg levodopa/hour)
  Other Names: ABT-SLV187; LCIG
Device: CADD-Legacy® 1400 ambulatory infusion pump
Device: PEG tube — percutaneous endoscopic gastrostomy tube
Device: J-tube — jejunal tube

SUMMARY:
The primary objective of this study is to measure the efficacy of ABT-SLV187 in subjects with advanced Parkinson's disease.

DETAILED DESCRIPTION:
The study was composed of a screening period followed by 2 sequential on-treatment periods, as follows:

* Screening Period (up to 28 days): determination of eligibility and discontinuation of antiparkinsonian disease medications other than levodopa-carbidopa immediate release (LC-oral) prior to nasojejunal (N-J) tube placement.
* N-J Test Period (2 to 14 days): first hospitalization period, Baseline assessments, placement of N-J tube, and optimization of levodopa-carbidopa intestinal gel (LCIG) treatment via N-J tube and infusion pump (participant was hospitalized for N-J tube placement but hospitalization was not required for entire duration of LCIG treatment optimization).
* PEG-J Period (12 weeks): second hospitalization period; placement of PEG-J tube; further optimization of LCIG treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria.
2. Subjects have 4 or 5 in modified Hohn and Yahr (H & Y) classification of disease severity at "Off" state determined by the UPDRS Part V at Screening Visit 1.
3. The subject's advanced Parkinson's disease must be levodopa-responsive as judged by the Investigator.
4. Subjects have had optimal treatment with available Parkinson's disease medication as defined by local standards of care and, based upon the judgment of the Investigator, and their symptoms are judged inadequately controlled on this optimized treatment. Optimized treatment is defined as the maximum therapeutic effect obtained with available anti-parkinsonian pharmacological therapy when no further improvement is expected regardless of any additional manipulations of levodopa and/or other anti parkinsonian medication; this will be based on the Investigator's best clinical judgment.
5. Presence of a recognizable "Off" and "On" state (motor fluctuations) as confirmed by UPDRS Part III (in both "On" and "Off" states), and by the Parkinson's Disease Diary© which must be observed and confirmed at Screening Visit 1.
6. Subjects must be experiencing a minimum of 3 hours per day of "Off" time, as estimated by the Investigator and supported by the UPDRS at Screening Visit 1 and the Parkinson's Disease Diaries at baseline. The "Off" time must occur during a continuous 16-hour interval, including the portion of the day during which the subject is awake the majority of the time (e.g., 5 AM to 9 PM, 7 AM to 11 PM).

Exclusion Criteria:

1. Parkinson's disease diagnosis is unclear or a suspicion of other parkinsonian syndromes exists, such as secondary Parkinsonism (caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), Parkinson's-plus syndromes (e.g., multiple system atrophy, progressive supranuclear palsy) or the other neurodegenerative diseases that might mimic the symptoms of Parkinson's disease .
2. Subjects who have undergone neurosurgery for the treatment of Parkinson's disease .
3. Current primary psychiatric diagnosis of acute psychotic disorder or other uncontrolled primary psychiatric diagnoses, (e.g., bipolar disorder or major depressive disorder per Diagnostic and Statistical Manual of Mental Disorders 4th edition, Text Revision (DSM-IV-TR) criteria.
4. Alzheimer's disease; or other significant cognitive impairment or dementia (defined as Mini-Mental State Examination (MMSE) total score < 24).
5. Subject has significant current suicidal ideation within the previous year as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) completed at Screening or any history of suicide attempts.
6. A low B12 level or low-normal B12 level (less than 300 pg/mL) with elevated methylmalonic acid (MMA). Note: Abnormal Vitamin B12 of questionable clinical significance (i.e., indeterminate or low normal results) prior to or at Screening Visit 2 require appropriate interpretation in conjunction with MMA and homocysteine laboratory values prior to proceeding further into the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masayoshi Yanagawa, PhD, Study Director — AbbVie Japan

REFERENCES:
- [Result] Murata M, Mihara M, Hasegawa K, Jeon B, Tsai CH, Nishikawa N, Oeda T, Yokoyama M, Robieson WZ, Ryman D, Eaton S, Chatamra K, Benesh J. Efficacy and safety of levodopa-carbidopa intestinal gel from a study in Japanese, Taiwanese, and Korean advanced Parkinson's disease patients. NPJ Parkinsons Dis. 2016 Nov 3;2:16020. doi: 10.1038/npjparkd.2016.20. eCollection 2016. PMID 28725701
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 participants were enrolled and had undergone the N-J placement procedure and were included in the Safety Analysis Set; 1 participant did not have at least 1 post-PEG efficacy assessment and was excluded from the Full Analysis Set (FAS), which consisted of 30 participants.
Period: Overall Study
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Started | 31
Completed | 28
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects who had undergone the N-J placement procedure.
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 12
Duration of Parkinson's Disease Since Initial Diagnosis [Mean (Standard Deviation); unit: years] | 12.4 (5.08)

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Normalized "Off" Time: Change From Baseline To The Final PEG-J Visit
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Negative change from baseline for "off" time indicates improvement.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the Full Analysis Set (FAS; all enrolled participants who received at least 1 dose of LCIG infusion during the PEG-J Period and had data for baseline and at least 1 post-PEG-J efficacy assessment) with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
hours
  Baseline | 7.37 (2.263)
  Last PEG-J visit | 2.72 (2.320)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -4.64, 95% CI 2-sided [-5.78 to -3.50]

2. Secondary Outcome: Average Daily Normalized "On" Time Without Troublesome Dyskinesia: Change From Baseline To The Final PEG-J Visit
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Positive change from baseline for "on" time indicates improvement.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
hours
  Baseline | 7.52 (2.505)
  Last PEG-J visit | 13.10 (2.453)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = 5.58, 95% CI 2-sided [4.21 to 6.95]

3. Secondary Outcome: Parkinson's Disease Questionnaire (PDQ-39) Summary Index: Change From Baseline To The Final PEG-J Visit
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The PDQ-39 Summary Index is the sum of all answers divided by the highest score possible (i.e. number of answers multiplied by 4) which is multiplied by 100 to put the score on a 0-100 scale. Higher scores are associated with more severe symptoms.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 35.5 (13.75)
  Last PEG-J visit | 23.5 (13.59)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -12.0, 95% CI 2-sided [-16.3 to -7.7]

4. Secondary Outcome: Clinical Global Impression - Change (CGI-I) Score at the Final PEG-J Visit
Description: The CGI-I is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-I ratings are as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: Final PEG-J Visit (up to week 12)
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
units on a scale | 1.9 (0.77)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); The p-value is based on a one-sample Wilcoxon signed-rank test with the hypothesis of no change (score = 4); Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean change from score = 4 = -2.1, Standard Deviation 0.77

5. Secondary Outcome: Patient Global Impression of Change (PGI-C) Score at the Final PEG-J Visit
Description: The PGI-C is a 7-point response scale. The subjects were to rate their change in status from Screening Visit 1 using the following 7-point scale: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse. The responses of "Minimally improved," "Much improved," and "Very much improved" on the PGI-C were used to define responders.
Time Frame: Final PEG-J Visit (up to week 12)
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
units on a scale | 2.0 (0.94)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); The p-value is based on a one-sample Wilcoxon signed-rank test with the hypothesis of no change (score = 4); Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean change from score = 4 = -2.0, Standard Deviation 0.94

6. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score: Change From Baseline To The Final PEG-J Visit
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 9.4 (6.63)
  Last PEG-J visit | 7.6 (6.93)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.101, One-sample t-test, 2-sided; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.0 to 0.4]

7. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part IIl Score: Change From Baseline To The Final PEG-J Visit
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part III score is the sum of the 27 answers provided to the 14 Part III questions, each of which are measured on a 5-point scale (0-4). The Part III score ranges from 0-108 and higher scores are associated with more disability.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 16.5 (9.70)
  Final PEG-J visit | 14.3 (11.30)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.182, One-sample t-test, 2-sided; Mean Difference (Net) = -2.1, 95% CI 2-sided [-5.3 to 1.1]

8. Secondary Outcome: Average Daily Normalized "On" Time With Troublesome Dyskinesia: Change From Baseline To The Final PEG-J Visit
Description: as for outcome 2
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
hours
  Baseline | 1.12 (2.311)
  Last PEG-J visit | 0.12 (0.394)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.032, One-sample t-test, 2-sided; Mean Difference (Net) = -1.00, 95% CI 2-sided [-1.90 to -0.09]

9. Secondary Outcome: Parkinson's Disease Questionnaire (PDQ-39) Mobility, Emotional Well-Being, Stigma, Social Support, Cognition, Communication, and Bodily Discomfort Domain Scores: Change From Baseline To The Final PEG-J Visit
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items (each question answered on a 5-point scale) addressing 8 domains of health in Parkinson's disease patients: Mobility (e.g., fear of falling when walking) includes 10 questions; Emotional Well-being (e.g., feelings of isolation) includes 6 questions; Stigma (e.g., social embarrassment) includes 4 questions; Social Support includes 3 questions; Cognition includes 4 questions; Communication includes 3 questions; and Bodily Discomfort includes 3 questions. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Mobility Domain-Baseline | 55.7 (19.46)
  Mobility Domain-Last PEG-J visit | 36.5 (22.49)
  Emotional Well-Being Domain-Baseline | 30.8 (19.13)
  Emotional Well-Being Domain-Last PEG-J visit | 24.3 (18.02)
  Stigma Domain-Baseline | 20.6 (22.21)
  Stigma Domain-Last PEG-J visit | 13.1 (20.78)
  Social Support Domain-Baseline | 16.1 (18.69)
  Social Support Domain-Last PEG-J visit | 14.6 (21.35)
  Cognition Domain-Baseline | 28.5 (19.26)
  Cognition Domain-Last PEG-J visit | 14.6 (13.16)
  Communication Domain-Baseline | 13.3 (14.62)
  Communication Domain-Last PEG-J visit | 14.4 (16.94)
  Bodily Discomfort Domain-Baseline | 35.0 (21.60)
  Bodily Discomfort Domain-Last PEG-J visit | 17.2 (14.83)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Mobility Domain analysis; Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -19.2, 95% CI 2-sided [-27.8 to -10.6]
Statistical Analysis 2: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Emotional Well-Being Domain analysis; Test type: Superiority or Other; p = 0.059, One-sample t-test, 2-sided; Mean Difference (Net) = -6.5, 95% CI 2-sided [-13.3 to 0.3]
Statistical Analysis 3: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Stigma Domain analysis; Test type: Superiority or Other; p = 0.070, One-sample t-test, 2-sided; Mean Difference (Net) = -7.5, 95% CI 2-sided [-15.6 to 0.6]
Statistical Analysis 4: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Social Support Domain analysis; Test type: Superiority or Other; p = 0.591, One-sample t-test, 2-sided; Mean Difference (Net) = -1.5, 95% CI 2-sided [-7.3 to 4.2]
Statistical Analysis 5: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Cognition Domain analysis; Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -14.0, 95% CI 2-sided [-20.7 to -7.3]
Statistical Analysis 6: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Communication Domain analysis; Test type: Superiority or Other; p = 0.670, One-sample t-test, 2-sided; Mean Difference (Net) = 1.1, 95% CI 2-sided [-4.2 to 6.4]
Statistical Analysis 7: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Bodily Discomfort Domain analysis; Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -17.8, 95% CI 2-sided [-25.2 to -10.3]

10. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total Score: Change From Baseline To The Final PEG-J Visit
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The total score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale. The total score will range from 0 to176, with 176 representing the worst (total) disability, and 0 representing no disability.
Time Frame: Baseline and Final PEG-J Visit (up to Week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 27.7 (15.53)
  Last PEG-J visit | 22.9 (17.53)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.056, One-sample t-test, 2-sided; Mean Difference (Net) = -4.8, 95% CI 2-sided [-9.8 to 0.1]

11. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score: Change From Baseline To The Final PEG-J Visit
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part I Score is the sum of the answers to the 4 questions that comprise Part I, each of which are measured on a 5-point scale (0-4). The Part I score ranges from 0 to 16 and higher scores are associated with more disability.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 1.8 (2.02)
  Last PEG-J visit | 0.9 (0.91)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p = 0.011, One-sample t-test, 2-sided; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.6 to -0.2]

12. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Score: Change From Baseline To The Final PEG-J Visit
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part IV Score is the sum of the answers to the 11 questions that comprise Part IV, each of which are measured on a 5-point scale (0-4) or a 2-point scale (0 or 1). The Part IV score ranges from 0 to 23 and higher scores are associated with more disability.
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 30
units on a scale
  Baseline | 8.7 (3.15)
  Last PEG-J visit | 5.5 (3.08)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -3.2, 95% CI 2-sided [-4.4 to -1.9]

13. Secondary Outcome: Average Daily Normalized "Off" Time Excluding Subjects Who Did Not Receive LCIG During the Entire PEG-J Period: Change From Baseline To The Final PEG-J Visit
Description: as for outcome 1
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 28
hours
  Baseline | 7.32 (2.290)
  Last PEG-J visit | 2.67 (2.341)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -4.65, 95% CI 2-sided [-5.83 to -3.47]

14. Secondary Outcome: Average Daily Normalized "Off" Time Including All PD Diaries Regardless if They Were Completed After the Subject Had Used a Concomitant Anti-Parkinsonian Medication: Change From Baseline To The Final PEG-J Visit
Description: as for outcome 1
Time Frame: Baseline (end of screening period) and Final PEG-J Visit (up to week 12)
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
hours
  Baseline | 7.37 (2.263)
  Last PEG-J visit | 2.78 (2.382)
Statistical Analysis 1: Comparison: Levodopa-Carbidopa Intestinal Gel (LCIG); Test type: Superiority or Other; p < 0.001, One-sample t-test, 2-sided; Mean Difference (Net) = -4.58, 95% CI 2-sided [-5.73 to -3.44]

15. Secondary Outcome: Average Daily Normalized "Off" Time at Baseline and Each Visit: Change From Baseline To The Final PEG-J Visit
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. n= the number of participants with available data at each time point.
Time Frame: Baseline (end of screening period) and Weeks 2, 4, 6, 8, 10, and 12
Population: All participants in the FAS with available data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 29
hours
  Baseline (n=29) | 7.37 (2.263)
  Week 2 (n=29) | 3.17 (2.365)
  Week 4 (n=29) | 3.68 (3.077)
  Week 6 (n=29) | 2.61 (2.318)
  Week 8 (n=27) | 2.77 (2.324)
  Week 10 (n=27) | 2.47 (2.210)
  Week 12 (n=27) | 2.45 (2.094)

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent AEs (TEAEs) are defined as any event that began or worsened in severity after N-J placement. The investigator assessed the relationship of each event to the use of study drug as Reasonable Possibility or No Reasonable Possibility.
  For more details on adverse events please see the AE section below.
Time Frame: From N-J placement to the end of study or early termination of treatment, including the removal of PEG-J (up to 17 weeks), plus 30 days.
Population: Safety Analysis Set: All subjects who had undergone the N-J placement procedure.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 31
participants
  Any TEAE | 31
  Any TEAE at least possibly related to LCIG | 0
  Any TEAE at least possibly related to LCIG System | 30
  Any severe TEAE | 2
  Any SAE | 4
  Any TEAE Leading to Discontinuation of Study | 1
  Death | 1
  Death related to AE | 1

17. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Parameters
Description: Terms abbreviated in the table include supine systolic blood pressure (SuSBP), standing systolic blood pressure (StSBP), orthostatic systolic blood pressure (OSBP), supine diastolic blood pressure (SuDBP), standing diastolic blood pressure (StDBP), orthostatic diastolic blood pressure (ODBP), supine pulse (SuP) in beats per minute (bpm), standing pulse (StP), body temperature (Temp), and baseline (BL). Increase and decrease are signified by ↑ and ↓, respectively.
Time Frame: From Baseline (end of screening period) to Final PEG-J Visit (up to week 12)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 31
participants
  SuSBP <=90 and >30 mm Hg ↓ from BL | 3
  SuSBP >=180 and >40 mm Hg ↑ from BL | 1
  StSBP <=90 and >30 mm Hg ↓ from BL | 3
  StSBP >=180 and >40 mm Hg ↑ from BL | 1
  OSBP: ↓ >=30 mm Hg Supine to Standing | 8
  SuDBP <=50 and >30 mm Hg ↓ from BL | 1
  SuDBP >=105 and >30 mm Hg ↑ from BL | 1
  StDBP <=50 and >30 mm Hg ↓ from BL | 3
  StDBP >=105 and >30 mm Hg ↑ from BL | 3
  ODBP: ↓ >=20 mm Hg Supine to Standing | 11
  SuP <=50 and >30 bpm ↓ from BL | 0
  SuP >=120 and >30 bpm ↑ from BL | 0
  StP <=50 and >30 bpm ↓ from BL | 0
  StP >=120 and >30 bpm ↑ from BL | 0
  Weight <=7% ↓ from BL | 8
  Weight >=7% ↑ from BL | 2

18. Secondary Outcome: Number of Participants With Potentially Clinically Significant Values for Hematology Parameters
Description: Terms abbreviated in the table include females (f), males (m), and femtoliters (fL).
Time Frame: From Baseline (end of screening period) to Final PEG-J Visit (up to week 12)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 31
participants
  Haemoglobin <90 g/L (f); <100 g/L (m) | 1
  Haematocrit <30% (f); <34% (m) | 2
  Red Blood Cells <2.0 10^12/L (f); <2.5 10^12/L (m) | 0
  Platelet Count <95 10^9/L | 1
  Platelet Count >700 10^9/L | 0
  White Blood Cells <2.8 10^9/L | 0
  White Blood Cells >16.0 10^9/L | 1
  Lymphocytes >80% | 0
  Monocytes >30% | 0
  Eosinophils >10% | 1
  Mean Corpuscular Volume <60 fL | 0
  Mean Corpuscular Volume >120 fL | 0

19. Secondary Outcome: Number of Participants With Potentially Clinically Significant Values for Clinical Chemistry Parameters
Description: Terms abbreviated in the table include upper limit of normal (ULN), male (m), and female (f).
Time Frame: From Baseline (end of screening period) to Final PEG-J Visit (up to week 12)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 31
participants
  Alanine Aminotransferase >3xULN | 1
  Aspartate Aminotransferase >3xULN | 1
  Gamma-glutamyl Transferase >3x ULN | 0
  Alkaline Phosphatase >400 U/L | 0
  Total Bilirubin >2xULN | 0
  Creatine Phosphokinase >3x ULN | 0
  Creatinine >177 µmol/L | 0
  Blood Urea Nitrogen >10.8 mmol/L | 2
  Uric Acid>500µmol/L(f);>590µmol/L(m) | 0
  Calcium <1.75 mmol/L | 0
  Calcium >3.0 mmol/L | 0
  Sodium <126 mmol/L | 0
  Sodium >156 mmol/L | 0
  Potassium <3.0 mmol/L | 1
  Potassium >6.0 mmol/L | 0
  Non-fasting Glucose <2.78 mmol/L | 1
  Non-fasting Glucose >16.0 mmol/L | 1
  Albumin <25 g/L | 1
  Albumin >70 g/L | 0
  Total Protein <45 g/L | 0
  Cholesterol >12.9 mmol/L | 0
  Triglycerides >5.6 mmol/L | 0
  Lactate dehydrogenase >3x ULN | 0

20. Secondary Outcome: Number of Participants With Potentially Clinically Significant Values for 12-lead Electrocardiogram (ECG)
Description: Terms abbreviated in the table include heart rate (HR) in beats per minute (bpm), PR interval (PRI), QT interval corrected for heart rate using Bazett's formula (QTcB), QT interval corrected for heart rate using Fridericia's formula (QTcF), and baseline (BL). Increase and decrease are signified by ↑ and ↓, respectively. n = the number of participants with available data at each time point.
Time Frame: From Baseline (end of screening period) to Final PEG-J Visit (up to week 12)
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Number analyzed (Participants) | 31
participants
  HR <=50 and >30 bpm ↓ from BL (n=31) | 0
  HR >=120 and >30 bpm ↑ from BL (n=31) | 0
  PR Interval <120 msec (n=30) | 0
  PR Interval >220 msec (n=30) | 1
  QTcB Interval >480 msec (n=31) | 1
  QTcB Interval >60 msec ↑ from BL (n=31) | 1
  QTcF Interval >480 msec (n=31) | 0
  QTcF Interval >60 msec ↑ from BL (n=31) | 1

21. Other Pre Specified Outcome: Neurological Examination
Description: Any abnormal findings are recorded as an adverse event after the first study drug administration; please see the AE section below. Further analysis for neurological examination findings was not performed per protocol.
Time Frame: From Baseline (end of screening period) to Final PEG-J Visit (up to week 12)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Physical Examination
Description: Any abnormal findings are recorded as an adverse event after the first study drug administration; please see the AE section below. Further analysis for physical examination findings was not performed per protocol.
Time Frame: From Baseline (end of screening period) to Final PEG-J Visit (up to week 12)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study enrollment to the end of study or early termination of treatment, including the removal of PEG-J (up to 17 weeks), plus 30 days.
Description: Serious AEs and treatment-emergent AEs are presented. Treatment-emergent AEs were defined as AEs that began or worsened from date of the N-J placement to 30 days after device removal or until the first dose of extension study drug for those who chose to continue LCIG treatment.
Arm/Group | Levodopa-Carbidopa Intestinal Gel (LCIG)
Serious Adverse Events (participants affected / at risk) | 4/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (LCIG) (N=31)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1
MELAENA (Gastrointestinal disorders) | 1
DEVICE DISLOCATION (General disorders) | 1
DEVICE KINK (General disorders) | 1
SEPSIS (Infections and infestations) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levodopa-Carbidopa Intestinal Gel (LCIG) (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 3
CARDIAC VALVE DISEASE (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
VITREOUS FLOATERS (Eye disorders) | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 6
DENTAL CARIES (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 6
DRY MOUTH (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 1
TOOTHACHE (Gastrointestinal disorders) | 2
CATHETER SITE PAIN (General disorders) | 1
CATHETER SITE PRURITUS (General disorders) | 1
CHEST DISCOMFORT (General disorders) | 1
CHEST PAIN (General disorders) | 1
COMPLICATION OF DEVICE INSERTION (General disorders) | 2
PYREXIA (General disorders) | 2
ALVEOLAR OSTEITIS (Infections and infestations) | 1
BODY TINEA (Infections and infestations) | 1
CATHETER SITE INFECTION (Infections and infestations) | 1
INCISION SITE CELLULITIS (Infections and infestations) | 1
INCISION SITE INFECTION (Infections and infestations) | 1
NASOPHARYNGITIS (Infections and infestations) | 6
RHINITIS (Infections and infestations) | 1
SIALOADENITIS (Infections and infestations) | 1
STOMA SITE CELLULITIS (Infections and infestations) | 1
STOMA SITE INFECTION (Infections and infestations) | 2
TINEA PEDIS (Infections and infestations) | 3
CONTUSION (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 6
INCISION SITE DERMATITIS (Injury, poisoning and procedural complications) | 1
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 4
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 13
INCISION SITE RASH (Injury, poisoning and procedural complications) | 2
LACERATION (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 5
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
SCRATCH (Injury, poisoning and procedural complications) | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 1
STOMA SITE ERYTHEMA (Injury, poisoning and procedural complications) | 1
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 2
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1
BLOOD HOMOCYSTEINE INCREASED (Investigations) | 5
BLOOD PRESSURE DECREASED (Investigations) | 2
BLOOD PRESSURE INCREASED (Investigations) | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
POSTURE ABNORMAL (Musculoskeletal and connective tissue disorders) | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1
DYSKINESIA (Nervous system disorders) | 5
DYSTONIA (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 2
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1
MIGRAINE (Nervous system disorders) | 1
RADICULOPATHY (Nervous system disorders) | 1
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1
AGITATION (Psychiatric disorders) | 1
ANXIETY (Psychiatric disorders) | 3
HEAD BANGING (Psychiatric disorders) | 1
ILLUSION (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 2
NIGHTMARE (Psychiatric disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1
ACNE (Skin and subcutaneous tissue disorders) | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 2
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 10
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
PETECHIAE (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1
HYPERTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.